CLINICAL TRIAL: NCT01272947
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Diclofenac Sodium Topical Gel (DSG) 1% Applied Four Times Daily in Subjects With Acute Blunt Soft Tissue Injuries/Contusions of the Limbs
Brief Title: Efficacy and Safety of Diclofenac Sodium Topical Gel 1% Applied Four Times Daily in Subjects With Acute Blunt Trauma Injuries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VOSG-P-319
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2012-12

CONDITIONS: Acute Blunt Soft Tissue Injuries/Contusions
Keywords: Blunt soft tissue injury/contusion
MeSH Terms: conditions — Contusions | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac sodium topical gel 1% (Experimental)
  Interventions: Drug: Diclofenac sodium
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diclofenac sodium — Topical gel 1%- 4 times daily
  Arms: Diclofenac sodium topical gel 1%
Other: Placebo — Topical gel - 4 times daily
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of DSG 1% compared with placebo applied four times a day in subjects with acute blunt soft tissue injuries/contusions of the limbs

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and over.
* Fresh impact injury (blunt, traumatic soft tissue injury or contusion) of the upper or the lower limbs, not requiring admittance to hospital, meeting baseline pain intensity level.Anticipated time between injury and treatment must be less than 3 hours.

Exclusion Criteria:

* Pain medication was taken within the 6 hours that precede randomization.Any physical impairment that would influence the study's efficacy evaluations, in particular POM such as: peripheral or central neurological disease, significant back pain; in case of acute blunt soft tissue injuries of the lower limbs: symptomatic osteoarthritis of the hips, knees, or feet, or any other painful conditions of the lower extremities (e.g., painful nail, wound, corn, or wart), in case of acute blunt soft tissue injuries of the upper limbs: no painful conditions of the upper extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - NCH investigative site, Brühl
  - NCH investigative site, Butzbach
  - NCH investigative site, Cologne
  - NCH investigative site, Essen
  - NCH investigative site, Gilching
  - NCH investigative site, Munich

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Started | 104 | 100
Completed | 102 | 98
Not Completed | 2 | 2
Not completed — Abnormal Laboratory Value | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo | Total
Number analyzed (Participants) | 104 | 100 | 204
Age Continuous [Mean (Standard Deviation); unit: years]
  Unit : years | 29.4 (9.6) | 31.4 (12.1) | 30.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 48 | 103
  Male | 49 | 52 | 101
Region of Enrollment [Number; unit: participants]
  Germany | 104 | 100 | 204

OUTCOME MEASURES:

1. Primary Outcome: Pain on Movement
Description: Visual analog scale (VAS) assessed on a 100 mm scale with anchors at 0= "No pain" and 100= "Extreme pain"
Time Frame: VAS Score at 24 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 104 | 100
mm | 33.1 (21.4) | 65.4 (16.9)

2. Secondary Outcome: Onset of Pain Relief
Description: Onset of perceptible pain relief.
Time Frame: From randomization to end of day 1
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 104 | 100
Hours | 2 [1 to 4] | NA [4.9 to NA] — The median time was not reached in the placebo group.

ADVERSE EVENTS:
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/100
Other Adverse Events (participants affected / at risk) | 2/104 | 4/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Topical Gel 1% (N=104) | Placebo (N=100)
Infections and Infestations (Infections and infestations) | 2 (2) | 3 (3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the Principal Investigator